CLINICAL TRIAL: NCT05389462
Title: A Phase 1b, Open-Label, Dose-Escalation and Dose-Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of Mipasetamab Uzoptirine (ADCT-601) Monotherapy and in Combination With Other Anti-Cancer Therapies in Patients With Selected Advanced Solid Tumors
Brief Title: A Study of Mipasetamab Uzoptirine (ADCT-601) in Participants With Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decided to halt further development of ADCT-601
Sponsor: ADC Therapeutics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADCT-601-102; 2021-005566-18 (EudraCT Number)
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced solid tumors; Mipasetamab uzoptirine; ADCT-601; Sarcoma; Gemcitabine; AXL; Pancreatic cancer; NSCLC
MeSH Terms: conditions — Sarcoma; Pancreatic Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Dose Escalation, ADCT-601 Combination Therapy (Experimental): In Part 1 (dose escalation), participants with selected sarcoma indications will receive escalating doses of ADCT-601 in combination with gemcitabine.
  Interventions: Drug: ADCT-601; Drug: Gemcitabine
- Part 1: Dose Escalation, ADCT-601 Monotherapy (Experimental): In Part 1 (dose escalation), participants with sarcoma indications (regardless of AXL gene amplification status), non-small-cell lung cancer (NSCLC) (regardless of AXL gene amplification status), and solid tumors with AXL gene amplification, will receive ADCT-601 monotherapy.
  Interventions: Drug: ADCT-601
- Part 2: Dose Expansion, ADCT-601 Combination Therapy (Experimental): In Part 2 (dose expansion), participants with selected sarcoma indications will receive ADCT-601 in combination with gemcitabine.
  Participants will be split into 3 cohorts:
  Cohorts 5 and 6: Sarcoma indications.
  Cohort 7: Pancreatic cancer.
  Interventions: Drug: ADCT-601; Drug: Gemcitabine
- Part 2: Dose Expansion, ADCT-601 Monotherapy (Experimental): In Part 2 (dose expansion), participants with a selected indication will receive ADCT-601 monotherapy.
  Participants will be split into cohorts:
  Cohort 1: Soft tissue sarcoma (STS).
  Cohort 2: Pancreatic adenocarcinoma (PAAD).
  Cohort 3: NSCLC.
  Cohort 4: Solid tumors with known AXL expression.
  Interventions: Drug: ADCT-601

INTERVENTIONS:
Drug: ADCT-601 — Intravenous (IV) infusion
  Other Names: Mipasetamab uzoptirine
Drug: Gemcitabine — Intravenous (IV) infusion
  Arms: Part 1: Dose Escalation, ADCT-601 Combination Therapy; Part 2: Dose Expansion, ADCT-601 Combination Therapy

SUMMARY:
The primary objective of this study is to identify the recommended phase 2 dose (RP2D) and/or the maximum tolerated dose (MTD), and characterize the safety and tolerability of ADCT-601 monotherapy and in combination with gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participant aged 18 years or older.
2. Pathologic diagnosis of solid tumor malignancy that is locally advanced or metastatic at time of screening:

   Part 1:
   1. Combination therapy arms: Selected sarcoma indications from the following 2 separate categories.

      * Soft tissue sarcoma: leiomyosarcoma, liposarcoma, undifferentiated pleomorphic sarcoma (UPS; covering malignant fibrous histiocytoma) and synovial sarcoma.
      * Bone sarcoma: Ewing's sarcoma (including extraskeletal), osteosarcoma, and chondrosarcoma.
   2. Monotherapy arms:

      * Sarcoma indications (including those listed for combination therapy arms) regardless of AXL gene amplification status.
      * NSCLC regardless of AXL gene amplification status.
      * Solid tumors (lymphomas participants are excluded) with known AXL gene amplification.

   Part 2:
   1. Combination therapy arms: Sarcoma indications and PAAD.
   2. Monotherapy arms: PAAD, NSCLC and solid tumors with AXL expression.
3. Participants who are refractory to or intolerant to available standard therapy(ies) known to provide clinical benefit for their condition per Investigator judgment.
4. Participants with measurable disease as determined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1.
6. PAAD only: Royal Marsden Hospital Prognostic Score 0 - 1.

Exclusion Criteria:

1. History of recent infection requiring intravenous (IV) antibiotics, IV antiviral, or IV antifungal treatment within 4 weeks of Cycle 1 Day 1 (C1D1).
2. Symptomatic central nervous system (CNS) metastases or evidence of leptomeningeal disease (brain magnetic resonance imaging [MRI] or previously documented cerebrospinal fluid [CSF] cytology). Previously treated asymptomatic CNS metastases are permitted provided that the last treatment (systemic anticancer therapy and/or local radiotherapy) was completed ≥4 weeks prior to Day 1 except usage of low dose of steroids on a taper (i.e., up to 10 mg prednisone or equivalent on Day 1 and consecutive days is permissible if being tapered down). Participants with discrete dural metastases are eligible.
3. Clinically significant third space fluid accumulation (i.e., ascites requiring drainage or any serosal effusion that is either requiring drainage or associated with shortness of breath).
4. Active diarrhea Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 or a medical condition associated with chronic diarrhea (such as irritable bowel syndrome, inflammatory bowel disease).
5. Use of any other experimental medication within 14 days prior to start of study drug (C1D1).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2025-04-17 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability as Assessed by Number of Participants with Adverse Events (AEs) | Up to approximately 2 years
  Adverse events (AEs) and serious adverse events (SAEs) are defined as any untoward medical occurrence in participants whether or not considered related to the investigational medicinal product. Any clinically significant changes in vital signs, laboratory values, 12-lead electrocardiogram (ECG) and Eastern Cooperative Oncology Group (ECOG) performance status results will be recorded as AEs and SAEs.
Number of Participants who Experience a Dose Limiting Toxicity (DLT) | Day 1 to Day 21
Number of Participants who Experience a Dose Interruption | Up to approximately 2 years
Number of Participants who Experience a Dose Reduction | Up to approximately 2 years

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to approximately 2 years
Duration of Response (DOR) | Up to approximately 2 years
Progression-Free Survival (PFS) | Up to approximately 2 years
Overall Survival (OS) | Up to approximately 2 years
Serum Concentration of ADCT-601 Total Antibody, Pyrrolobenzodiazepine (PBD)-Conjugated Antibody, and Unconjugated Warhead SG3199 | Day 1 up to approximately 2 years
Maximum Concentration (Cmax) of ADCT-601 Total Antibody, Pyrrolobenzodiazepine (PBD)-Conjugated Antibody, and Unconjugated Warhead SG3199 in Serum | Day 1 up to approximately 2 years
Time to Maximum Concentration (Tmax) of ADCT-601 Total Antibody, Pyrrolobenzodiazepine (PBD)-Conjugated Antibody, and Unconjugated Warhead SG3199 in Serum | Day 1 up to approximately 2 years
Area Under the Concentration-time Curve from Time Zero to the Last Quantifiable Concentration (AUClast) of ADCT-601 Total Antibody, Pyrrolobenzodiazepine (PBD)-Conjugated Antibody, and Unconjugated Warhead SG3199 in Serum | Day 1 up to approximately 2 years
Area Under the Concentration-time Curve from Time Zero to the End of the Dosing Interval (AUCtau) of ADCT-601 Total Antibody, Pyrrolobenzodiazepine (PBD)-Conjugated Antibody, and Unconjugated Warhead SG3199 in Serum | Day 1 up to approximately 2 years
Area Under the Concentration-time Curve from Time Zero to Infinity (AUCinf) of ADCT-601 Total Antibody, Pyrrolobenzodiazepine (PBD)-Conjugated Antibody, and Unconjugated Warhead SG3199 in Serum | Day 1 up to approximately 2 years
Apparent Terminal Elimination Half-life (T1/2) of ADCT-601 Total Antibody, Pyrrolobenzodiazepine (PBD)-Conjugated Antibody, and Unconjugated Warhead SG3199 in Serum | Day 1 up to approximately 2 years
Apparent Clearance (CL) of ADCT-601 Total Antibody, Pyrrolobenzodiazepine (PBD)-Conjugated Antibody, and Unconjugated Warhead SG3199 in Serum | Day 1 up to approximately 2 years
Apparent Steady-state Volume of Distribution (Vss) of ADCT-601 Total Antibody, Pyrrolobenzodiazepine (PBD)-Conjugated Antibody, and Unconjugated Warhead SG3199 in Serum | Day 1 up to approximately 2 years
Accumulation Index (AI) of ADCT-601 Total Antibody, Pyrrolobenzodiazepine (PBD)-Conjugated Antibody, and Unconjugated Warhead SG3199 in Serum | Day 1 up to approximately 2 years
Number of Participants With an Anti-drug Antibody (ADA) Response to ADCT-601 | Day 1 up to approximately 2 years
Number of Participants With Anti-drug Antibody (ADA) Titers to ADCT-601 | Day 1 up to approximately 2 years

CONTACTS AND LOCATIONS:
Locations (14):
- United States (6):
  - Sarcoma Oncology Research Center, Santa Monica, California
  - Stanford Cancer Center, Stanford Medicine at Stanford University, Stanford, California
  - University of IOWA, Iowa City, Iowa
  - Washington University School of Medicine, St Louis, Missouri
  - Sarah Cannon at University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Vanderbilt University Medical Center (VUMC) - Ingram Cancer Center, Nashville, Tennessee
- France (3):
  - Institut Bergonié, Bordeaux, Gironde
  - Institut Léon Bérard, Lyon
  - Centre Antoine Lacassagne, Nice
- Spain (3):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Madrid Sanchinarro, Madrid
- United Kingdom (2):
  - The Royal Marsden NHS Foundation Trust, London, England
  - The Christie NHS Foundation Trust, Manchester, England

IPD SHARING:
Plan to Share IPD: No